CLINICAL TRIAL: NCT02795910
Title: Integrated Primary Care for Diabetes and Cardiovascular Disease in Less Developed Countries: Pragmatic Trial of the Practical Approach to Care Kit
Brief Title: Integrated Primary Care for Diabetes and Cardiovascular Disease
Acronym: PACKBrazDCVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Santa Catarina Federal University (Other); University of Cape Town (Other); Federal University of Bahia (Other); Medical Research Council, South Africa (Other); University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACKBrazil2
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus; Hypertension; Heart Failure; Ischemic Heart Disease; Cerebrovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Heart Failure; Myocardial Ischemia; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Doctors and nurses in each clinic will receive printed copies of the patient management tool (PMT) and outreach education training. First trainers will be trained, then trainers will train groups of doctors and nurses at their workplaces, showing them how to use the guidelines, and using their own patients and clinical problems as examples. This outreach training is repeated several times in short sessions
  Interventions: Behavioral: Outreach education training
- Control (Active Comparator): Doctors and nurses in each clinic will receive printed copies of the patient management tool (PMT) but will receive no outreach education training.
  Interventions: Behavioral: No outreach education training

INTERVENTIONS:
Behavioral: Outreach education training — Printed copies of the patient management tool (PMT) and outreach education training
  Arms: Intervention
Behavioral: No outreach education training — Printed copies of the patient management tool (PMT) without outreach education training
  Arms: Control

SUMMARY:
This study will evaluate a complex intervention based on a patient management tool (PMT), combined with educational outreach to primary care doctors, nurses and other health workers, in the Brazilian city of Florianopolis. The intervention is aimed at improving the quality of primary health care and health outcomes, in adults with diabetes and cardiovascular disease (CVD). The effectiveness of the intervention will be assessed by randomly allocating 48 primary care clinics to receive the intervention or not, and comparing patient and clinic level endpoints that reflect the health and quality of care provided over the following year. About 11000 patients known to have been diagnosed with diabetes mellitus and 32000 with CVD (defined as having a diagnosis of hypertension, ischemic heart disease, heart failure or cerebrovascular disease) in participating clinics will be included in the study. About 7800 of them have diagnoses of both CVD and stroke. The primary endpoints will be 1. Number of participants in whom at least one of the following tests was recorded: body mass index, plasma glucose, serum cholesterol, electrocardiogram, and 2. in participants with a diagnosis of hypertension recorded previously, average systolic blood pressure recorded. Secondary endpoints will include the individual components of the composite scores, health measures (hospital admissions and deaths), and indicators of appropriate diagnosis of comorbid conditions such as depression. Eligible patients will be identified and outcomes measured using electronic medical records.

DETAILED DESCRIPTION:
Diabetes mellitus and cardiovascular disease (diabetes and CVD) place a heavy and growing burden on people living in low and middle income countries. Many of them could be healthier if their disease was accurately diagnosed and correctly treated, but many are not. Doctors and nurses working in primary health care clinic are best placed people to diagnose and treat, especially where local clinics are near and free. But this raises two questions: 1. How to ensure that diabetes and CVD get the priority they need in overloaded clinics? 2. How to ensure rational evidence-based diagnosis and prescribing for diabetes and CVD? The investigators have developed a way of improving primary health care for people who have long term health conditions. It is a patient management tool (PMT), that is, a printed manual of flowcharts taking doctors and nurses from symptoms to diagnoses to treatments, tests or referrals, with advice on how to make decisions along the way about diagnoses, tests, treatments and referrals. They are prompted to think of other diseases and health problems that might be undetected or neglected. The package also includes a method of training known as outreach education. First trainers are trained, then trainers train groups of doctors and nurses at their workplaces, showing them how to use the guidelines, and using their own patients and clinical problems as examples. This outreach training is repeated several times in short sessions. The investigators' research in Africa has shown that this approach can be effective, cost effective, feasible and sustainable. It has been rolled out throughout South Africa and other African countries. But it has have not yet been shown to be effective for diabetes and CVD. The investigators have also not tried or evaluate it in Latin American countries, which have different health systems, and have many more doctors providing primary health care. Now co-investigators in the Brazilian city of Florianopolis have decided to put this educational package in place throughout the city, and have agreed to do so as a randomised controlled trial. This will clearly show whether PACK Brazil is effective, cost effective and feasible under Brazilian conditions. The core of the research will be a randomised controlled trial. 48 primary care clinics in the city will be randomly chosen either 1) to get the whole package of patient management tool plus training, or 2) only to get the patient management tool (which is expected to will make little difference without training). The investigators will compare patients in these two groups of clinics to see the effects of the training. They will use the clinics' electronic medical records to identify about 32000 adults diagnosed with diabetes and CVD. After the training starts they will follow these patients up for a year, and assess whether they are being appropriately treated and tested. The primary endpoints will be 1. Number of participants in whom at least one of the following tests was recorded: body mass index, plasma glucose, serum cholesterol, electrocardiogram, and 2. in participants with a diagnosis of hypertension recorded previously, average systolic blood pressure recorded. Secondary endpoints will include frequency of tests, the number who have each type of test, diastolic blood pressure in participants with hypertension, serum glucose levels in participants with diabetes, prescription of indicated treatments and treatment intensification, health measures (hospital admissions and deaths), and indicators of diagnosis and treatment of comorbid conditions such as depression. Eligible patients will be identified and outcomes measured using electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 years and over in July 2016
* Diagnosis of hypertension (ICD-10 code I10-I15), ischaemic heart disease (ICD-10 code I20-I25), heart failure (ICD-10 code I50), cerebrovascular disease (ICD-10 code I60-I69), or diabetes mellitus (ICD-10 code E10-E14) ever recorded since January 1st 2010, and attended a participating clinic for any reason during the first year of the trial

Exclusion Criteria:

* None

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40577 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk and diabetes testing | During the first year of the trial
  Number of participants in whom at least one of the following tests was recorded: body mass index, plasma glucose, glycated hemoglobin (HbA1c), serum cholesterol, electrocardiogram.
Systolic blood pressure | During the first year of the trial
  In participants with a diagnosis of hypertension recorded previously, and with systolic blood pressure >140 mm Hg recorded during 12 months before start of follow up, average systolic blood pressure recorded

SECONDARY OUTCOMES:
Diastolic blood pressure | During the first year of the trial
  Number of tests for cardiovascular and diabetes risk factors (body mass index, plasma or skin prick glucose, serum cholesterol, electrocardiogram, chest X ray) recorded for each participant
Number of tests | During the first year of the trial
  Number of tests for cardiovascular and diabetes risk factors (body mass index, plasma or skin prick glucose, serum cholesterol, electrocardiogram, chest X ray) recorded for each participant
BMI measured | During the first year of the trial
  Number of participants who had body mass index recorded at least once
Cholesterol tested | During the first year of the trial
  Number of participants who had serum cholesterol recorded at least once
ECG tested | During the first year of the trial
  Number of participants who had electrocardiogram recorded at least once
Chest X ray tested | During the first year of the trial
  Number of participants who had chest X ray recorded at least once
Glucose tested | During the first year of the trial
  Number of participants who had plasma glucose recorded at least once
Simvastatin prescribed | During the first year of the trial
  Number of participants in whom simvastatin was prescribed for the first time
Simvastatin dose changed | During the first year of the trial
  Number of participants in whom dose of simvastatin was changed
Depression diagnosed | During the first year of the trial
  Number of participants in whom a diagnosis of depression (ICD-10 code F32-F34) was recorded for the first time
Antidepressant diagnosed | During the first year of the trial
  Number of participants in whom antidepressant medication (tricyclic and related antidepressants, selective serotonin re-uptake inhibitors, and monoamine oxidase inhibitors) was prescribed for the first time
Heart failure diagnosed | During the first year of the trial
  Number of participants in whom a diagnosis of heart failure (ICD-10 code I50) was recorded for the first time
Ischemic heart disease diagnosed | During the first year of the trial
  Number of participants in whom a diagnosis of heart failure (ICD-10 code I50) was recorded for the first time
Cerebrovascular disease diagnosed | During the first year of the trial
  Number of participants in whom a diagnosis of cerebrovascular disease (ICD-10 code I60-I69) was recorded for the first time
Angina referral | During the first year of the trial
  Number of participants referred to a hospital or specialist with a diagnosis of angina pectoris (ICD code I20)
Hospital admission for CVD | During the first year of the trial
  Number of participants admitted to hospital for ischemic heart disease, heart failure, hypertension, cerebrovascular disease or peripheral vascular disease (ICD code I73)
All cause mortality | During the first year of the trial
  Number of participants who died
Death from CVD | During the first year of the trial
  Number of participants who died and in whom ischemic heart disease, heart failure, hypertension, or cerebrovascular disease was recorded as an underlying cause of death
Any hypertension controlled | During the first year of the trial
  In participants with an average systolic blood pressure greater than 140 mm Hg, or an average diastolic blood pressure greater than 90 mm Hg, recorded during 12 months before enrolment, the number of participants with systolic blood pressure 140 mm Hg or less and with diastolic blood pressure 90 mm Hg or less
Severe hypertension controlled | During the first year of the trial
  In participants with an average systolic blood pressure greater than 150 mm Hg, or an average diastolic blood pressure greater than 100 mm Hg, recorded during 12 months before enrolment, the number of participants with systolic blood pressure 140 mm Hg or less and with diastolic blood pressure 90 mm Hg or less
Number of glucose tests | During the first year of the trial
  In participants with a diagnosis of diabetes, number of times plasma glucose or glycated hemoglobin (HbA1c) recorded
Glycated hemoglobin (HbA1c) | During the first year of the trial
  In participants with a diagnosis of diabetes, average glycated hemoglobin (HbA1c) level recorded
Heart failure treatment | During the first year of the trial
  In participants with a diagnosis of heart failure, the number of new prescriptions for furosemide, hydrochlorothiazide, enalapril or carvedilol
Increased hypertension treatment | During the first year of the trial
  In participants with a diagnosis of hypertension, the number of participants with a prescription for increased dose of hydrochlorothiazide, enalapril, amlodipine or propanalol
Ischemic heart disease treatment | During the first year of the trial
  In participants with a diagnosis of ischemic heart disease, then number of participants with a new prescription of angiotensin converting enzyme inhibitor, isosorbide dinitrate, propanalol, enalapril or losartan

CONTACTS AND LOCATIONS:
Overall Officials: Max Bachmann, MBChB PhD, Principal Investigator — University of East Anglia; Eric Bateman, MBChB MD, Principal Investigator — University of Cape Town; Rafael Stelmach, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Florianopolis City Health Department, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachmann MO, Bateman ED, Stelmach R, Cruz AA, Pacheco de Andrade M, Zonta R, Zepeda J, Natal S, Cornick R, Wattrus C, Anderson L, Lombard C, Fairall LR. Integrating primary care of chronic respiratory disease, cardiovascular disease and diabetes in Brazil: Practical Approach to Care Kit (PACK Brazil): study protocol for randomised controlled trials. J Thorac Dis. 2018 Jul;10(7):4667-4677. doi: 10.21037/jtd.2018.07.34. PMID 30174920